CLINICAL TRIAL: NCT05227196
Title: A Bioequivalence Study of Two Formulations of Oral Semaglutide in Healthy Participants
Brief Title: A Research Study Looking at the Comparability of 2 Different Forms of Oral Semaglutide in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4799
Record Dates: First submitted 2022-02-02; First posted 2022-02-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 Sequence 1 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide D Dose 2; Drug: Semaglutide D Dose 3; Drug: Semaglutide Dose 6
- Group 1 Sequence 2 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 3; Drug: Semaglutide Dose 4; Drug: Semaglutide Dose 5; Drug: Semaglutide Dose 6
- Group 2 Sequence 1 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide D Dose 2; Drug: Semaglutide Dose 4; Drug: Semaglutide Dose 5
- Group 2 Sequence 2 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide D Dose 2; Drug: Semaglutide Dose 4; Drug: Semaglutide Dose 5
- Group 3 Sequence 1 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide Dose 4
- Group 3 Sequence 2 (Experimental): Crossover arm
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide Dose 4

INTERVENTIONS:
Drug: Semaglutide D Dose 1 — Tablet given orally
  Arms: Group 1 Sequence 1; Group 2 Sequence 1; Group 2 Sequence 2; Group 3 Sequence 1; Group 3 Sequence 2
Drug: Semaglutide D Dose 2 — Tablet given orally
  Arms: Group 1 Sequence 1; Group 2 Sequence 1; Group 2 Sequence 2
Drug: Semaglutide D Dose 3 — Tablet given orally
  Arms: Group 1 Sequence 1; Group 1 Sequence 2
Drug: Semaglutide Dose 4 — Tablet given orally
  Arms: Group 1 Sequence 2; Group 2 Sequence 1; Group 2 Sequence 2; Group 3 Sequence 1; Group 3 Sequence 2
Drug: Semaglutide Dose 5 — Tablet given orally
  Arms: Group 1 Sequence 2; Group 2 Sequence 1; Group 2 Sequence 2
Drug: Semaglutide Dose 6 — Tablet given orally
  Arms: Group 1 Sequence 1; Group 1 Sequence 2

SUMMARY:
The aim of this study is to investigate the amount of the active ingredient and helping agent in the blood in two different tablet versions of Semaglutide. The study will consist of 3 groups and the treatment the participants will get is dependent on the group the participants will be enrolled in.

The participants in group 1 will receive treatment for 22 weeks, group 2 for 21 weeks and group 3 for 20 weeks.

The study will last up to 29 to 31 weeks for each participant. This includes a screening period (up to 4 weeks), a dose escalation period (up to 2 weeks), a treatment period (20 weeks) and a follow-up period (5 weeks after the last dose).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent. - Body mass index (BMI) between 21.0 and 32.0 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* HbA1c equal to or greater than 6.5 % (48 mmol/mol) at screening.
* Use of tobacco and nicotine products, defined as any of the below:
* Smoking more than 5 cigarettes or the equivalent per day
* Not willing to refrain from smoking and use of nicotine substitute products within 48 hours prior to and during the inpatient periods
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.
* History(a) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant(a).
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma(a).

  1. As declared by the participant or reported in the medical records

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 546 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,semaglutide,SS Area under the semaglutide plasma concentration-time curve during a dosing interval at steady state (SS) | 24 hours after the dosing of oral semaglutide on days 35/42/49, 70/77/84, 105/112/119 and 140/147/154.
  h∙nmol/L
Cmax,0-24h.semaglutide,SS Maximum semaglutide plasma concentration at steady state | 24 hours after the dosing of oral semaglutide on days 35/42/49, 70/77/84, 105/112/119 and 140/147/154.
  nmol/L

SECONDARY OUTCOMES:
tmax,0-24h,semaglutide,SS Time to maximum semaglutide plasma contraction at steady state | 24 hours after the dosing of oral semaglutide on days 35/42/49, 70/77/84, 105/112/119 and 140/147/154.
  h
Ctau,24h,semaglutide,SS Semaglutide plasma concentration 24 hours after last dose at steady state | 24 hours after the dosing of oral semaglutide on days 35/42/49, 70/77/84, 105/112/119 and 140/147/154.
  nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept. 2834), Study Director — Novo Nordisk A/S
Locations (3):
- United States (2):
  - Altasciences Clinical LA, Inc., Cypress, California
  - Altasciences Clinical Kansas, Inc., Overland Park, Kansas
- Altasciences Company Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Nielsen MS, Brondsted L, Kankam M, Morelli G, Nguyen D, Skjoth TV, Patted UR, van Hout M. A Bioequivalence Study of Two Formulations of Oral Semaglutide in Healthy Participants. Diabetes Ther. 2025 Feb;16(2):269-287. doi: 10.1007/s13300-024-01674-8. Epub 2024 Dec 21. PMID 39708086